CLINICAL TRIAL: NCT00834847
Title: A Relative Bioavailability Food Challenge Study of Pravastatin Sodium 40 mg Tablets
Brief Title: Pravastatin Sodium 40 mg Tablets Food Challenge Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B006512
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pravastatin fast (Experimental): Test product under fasting conditions dosed in first period followed by either test or reference product dosed under fed conditions in second and third periods
  Interventions: Drug: pravastatin
- Pravastatin (Experimental): Test product under fed conditions dosed in first period followed by either test product dosed under fasting conditions or reference product dosed under fed conditions in second and third periods
  Interventions: Drug: pravastatin
- Pravachol® (Active Comparator): Reference product under fed conditions dosed in first period followed by test product dosed under either fed or fasted conditions in second and third periods
  Interventions: Drug: Pravachol®

INTERVENTIONS:
Drug: pravastatin — 40 mg tablet
  Arms: Pravastatin; Pravastatin fast
Drug: Pravachol® — 40 mg Tablet
  Arms: Pravachol®

SUMMARY:
The objective of this study is to compare the relative bioavailability of pravastatin 40 mg tablets with that of Pravachol 40 mg tablets in healthy adult male subjects under non-fasting conditions. A second objective is to compare the difference in plasma levels after dosing the test formulation with and without food.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria

* Non-institutionalized subjects consisting of university students and members of the community at large.
* All subjects selected for this study will be males 18 to 45 (inclusive) years of age. Weight of the subjects shall not be more than 15% from the normal for height and body frame (Metropolitan Life, 1993, Height, Weight, Body Chart).
* Each subject shall be given a general physical examination within 21 days of initiation of the study. Such examination includes, but is not limited to, blood pressure, general observations, and history.

At the end of the study the subjects will have an exit evaluation consisting of interim history, global evaluation, and clinical laboratory measurements.

Adequate blood and urine samples should be obtained within 21 days before the beginning of the first period and at the end of the trial for clinical laboratory measurements.

Clinical laboratory measurements will include the following:

Hematology: hemoglobin, hematocrit, red blood cell count, platelets, and white blood cell count (with differential)

Clinical Chemistry: creatinine, BUN, glucose, SGOT, SGPT, bilirubin, and alkaline phosphatase

Urine Analysis: pH, specific gravity, protein, glucose, ketones, bilirubin, occult blood, and cells

HIV Screen: (pre-study only)

Hepatitis-B, C Screen: (pre-study only)

Drugs of Abuse Screen: (pre-study and at each dosing period check-in)

Subjects will be selected if all above are normal. Electrocardiograms of all participating subjects will be recorded before initiation of the study and filed with each subject's case report forms.

Exclusion Criteria

* Subjects with a history of chronic alcohol consumption, drug addiction, or serious gastrointestinal, renal, hepatic, or cardiovascular disease, tuberculosis, epilepsy, asthma, diabetes, psychosis or glaucoma will not be eligible for this study.
* Subjects whose clinical laboratory test values are greater than 20% outside the normal range may be retested. If the clinical values are outside the range on retesting the subject will not be eligible to participate in the study unless the clinical investigator deems the result to not be significant.
* Subjects who have a history of allergic responses to the class of drug being tested should be excluded from the study.
* Subjects who use tobacco in any form will not be eligible to participate in the study. Three months abstinence is required.
* All subjects will have urine samples assayed for the presence of drugs of abuse as part of the clinical laboratory screening procedures and at each dosing period check-in. Subjects found to have urine concentrations of any of the tested drugs will not be allowed to participate.
* Subjects should not have donated blood and/or plasma for at least thirty (30) days prior to the first dosing of the study.
* Subjects who have taken any investigational drug within thirty (30) days prior to the first dosing of the study will not be allowed to participate.
* Subjects who have been exposed to known hepatic enzyme inducing or inhibiting agents within (30) days prior to dosing will not be allowed to participate.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2000-08; Primary Completion 2000-09 (Actual); Study Completion 2000-09 (Actual)

PRIMARY OUTCOMES:
Cmax - Maximum Observed Concentration | Blood samples collected over 24 hour period
AUC0-inf - Area under the concentration-time curve from time zero to infinity (extrapolated) | Blood samples collected over 24 hour period
AUC0-t - Area under the concentration-time curve from time zero to time of last non-zero concentration (per participant) | Blood samples collected over 24 hour period

SECONDARY OUTCOMES:
Cmax - Comparison of the difference in plasma levels after dosing with test product under fasted and fed conditions | Blood samples collected over 24 hour period
AUC0-inf - Comparison of the difference in plasma levels after dosing with test product under fasted and fed conditions | Blood samples collected over 24 hour period
AUC0-t - Comparison of the difference in plasma levels after dosing with test product under fasted and fed conditions | Blood samples collected over 24 hour period

CONTACTS AND LOCATIONS:
Overall Officials: Dan Yeung, MD, Principal Investigator — Pharma Medica
Locations (1):
- Pharma Medica Research Inc., Toronto, Ontario, Canada